CLINICAL TRIAL: NCT03651336
Title: A Prospective, Open-label, Multicenter Clinical Follow-up Investigation of the ARGOS-01 and ARGOS-02 Patients to Assess the Long-term Safety and Performance of the ARGOS-IO Intraocular Pressure Sensor System in Subjects With Primary Open Angle Glaucoma (POAG)
Brief Title: Long-term Safety and Performance of the ARGOS-IO Intraocular Pressure Sensor System in Subjects With Primary Open Angle Glaucoma (POAG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Implandata Ophthalmic Products GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ARGOS-03; CIV-18-13-023284 (Other: EUDAMED)
Record Dates: First submitted 2018-08-20; First posted 2018-08-29 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Primary Open-angle Glaucoma
Keywords: POAG; Primary Open Angle Glaucoma; Cataract; Intraocular Pressure; Intraocular Pressure Sensor System; IOP; Self-monitoring of intraocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm longterm follow-up ARGOS-IO Sensor Pressure System (Other): The ARGOS-IO sensor was already implanted in a previous study as ARGOS-01 or ARGOS-02.
  Interventions: Device: ARGOS-IO Sensor Pressure System

INTERVENTIONS:
Device: ARGOS-IO Sensor Pressure System — The ARGOS-IO Pressure sensor have been additionally implanted during local routine working procedures for cataract surgery in Patients with Primary Open Angle Glaucoma (POAG) and indicated cataract surgery in previous studies ARGOS-01 and ARGOS-02
  Other Names: EYEMATE-IO

SUMMARY:
The purpose of this study is to evaluate the long-term safety and performance of the ARGOS-IO system in patients with Primary Open Angle Glaucoma (POAG)

DETAILED DESCRIPTION:
This study is a prospective open-label, multicenter study for clinical follow-up of the ARGOS-01 and ARGOS-02 patients.

From the ARGOS-01 to the ARGOS-02 study, some modifications were made to the form of the ARGOS-IO implant in consequence of the outcomes of the ARGOS-01 study.

Maximal 5 patients of the ARGOS-01 study and maximal 21 patients of the ARGOS-02 study will take part in this study.

The sensor was always implanted in one eye only which will be the study eye.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of the ARGOS-01 and ARGOS-02 study with an implanted ARGOS-IO pressure sensor.

Exclusion Criteria:

* N/A

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagen Thieme, Prof., Principal Investigator — Universitätsaugenklinik Magdeburg
Locations (4):
- Germany (4):
  - Klinik für Augenheilkunde, Uniklinik RWTH Aachen, Aachen
  - Universitäts-Augenklinik Bochum, Bochum
  - Universitätsaugenklinik Magdeburg, Magdeburg
  - Universitäts-Augenklinik Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mansouri K, Rao HL, Weinreb RN. Nyctohemeral effects of topical beta-adrenoceptor blocking agents measured with an intraocular telemetry sensor. Br J Ophthalmol. 2025 Apr 22;109(5):582-586. doi: 10.1136/bjo-2023-324760. PMID 39510809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from August 2018 to May 2019 in medical clinics.
Groups:
- ARGOS-IO System: ARGOS-IO Pressure sensor previously implanted during local routine working procedures for cataract surgery in Patients with Primary Open Angle Glaucoma (POAG) and indicated cataract surgery in the ARGOS-01 and ARGOS-02 studies.
  ARGOS-IO system: An active implantable intraocular pressure sensor to be implanted in the ciliary sulcus of the human eye, in combination with cataract surgery.
Period: Overall Study
Arm/Group | ARGOS-IO System
Started | 16
Completed | 12
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- ARGOS-IO System: In this prospective open-label, multicenter study for clinical follow-up of the ARGOS-01 and ARGOS-02 patients, 16 patients were enrolled. Goldmann applanation tonometry (GAT) measurements were compared with the sensors' IOP measurements and comprehensive ophthalmic examinations were performed at all follow-up visits (V01-V07) through 36 months.
Arm/Group | ARGOS-IO System
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 16

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Patients Experiencing a Device Related Serious Adverse Events (SADE) and Device Related Adverse Events (ADE)
Description: Number of patients experiencing a device related SAE (SADE) and device related complications (ADE) over the 36-months' clinical follow-up time.
Time Frame: Baseline visit to Day 1080 (V01 [Baseline visit] to V07)
Measure: Count of Participants; unit: Participants
Arm/Group | ARGOS-IO System
Number analyzed (Participants) | 16
Participants
  SADEs | 0
  ADEs | 0

2. Primary Outcome: Performance: Level of Agreement Between GAT and the ARGOS-IO System
Description: Level of Agreement between intraocular pressure (IOP) measurements made using GAT & the ARGOS-IO system (IOP in mmHg) following the Bland-Altman method.
Time Frame: Baseline visit to Day 1080 (V01 [Baseline visit] to V07)
Population: All available pairs of GAT and the ARGOS-IO System IOP measurements.
Measure: Mean (95% Confidence Interval); unit: mmHg
Units Other Than Participants: IOP measurement pairs
Arm/Group | ARGOS-IO System
Number analyzed (Participants) | 16
Number analyzed (IOP measurement pairs) | 212
mmHg | 1.4 [-5.2 to 7.9]

3. Primary Outcome: Performance: Device Malfunctions
Description: Incidence, nature and seriousness of observed device malfunctions / deficiencies (DDs)
Time Frame: Baseline visit to Day 1080 (V01 [Baseline visit] to V07)
Population: All device deficiencies.
Measure: Number; unit: DDs
Units Other Than Participants: DDs
Arm/Group | ARGOS-IO System
Number analyzed (Participants) | 7
Number analyzed (DDs) | 8
DDs
  Reader device (external handheld device) | 8
  ARGOS-IO sensor | 0

4. Secondary Outcome: Patient's Compliance in IOP Self-monitoring (Daily Self-measurements)
Description: The patients' compliance in IOP self-monitoring throughout the clinical follow-up study. Daily self-measurements with the ARGOS-IO sensor were to be done at least 4 times daily (morning, noon, afternoon, evening).
Time Frame: Baseline visit to Day 1080 (V01 [Baseline visit] to V07)
Population: All available ARGOS-IO measurements. Of the 16 patients, 3 patients were not included in the summarizing analysis for reasons related to early withdrawal from the study and dementia, hence the 13 participants analyzed.
Measure: Mean (Standard Deviation); unit: percentage of daily self-measurements
Arm/Group | ARGOS-IO System
Number analyzed (Participants) | 13
percentage of daily self-measurements | 79 (29)

5. Secondary Outcome: Patient's Compliance in IOP Self-monitoring (Self-measurement Sequences / Day)
Description: as for outcome 4
Time Frame: Baseline visit to Day 1080 (V01 [Baseline visit] to V07)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: number of self-measurement sequences/day
Arm/Group | ARGOS-IO System
Number analyzed (Participants) | 13
number of self-measurement sequences/day | 3.4 (0.9)

ADVERSE EVENTS:
Time Frame: Evaluation over 36 months' follow-up period.
Description: SAE Definition
  That meets any of the following criteria of a serious adverse event:
  * Resulted in death, permanent damage or disability or a congenital anomaly
  * Was life threatening
  * Required hospitalization
Groups:
- ARGOS-IO System: A total of 16 patients from the ARGOS-01 and ARGOS-02 studies were enrolled in this open-label, multicenter study for clinical follow-up. Throughout the 36 months' clinical follow-up, the patients returned for 8 follow-up visits (V01-V07) consisting of comprehensive ophthalmic examinations as well as IOP measurements with the ARGOS-IO system and GAT.
Arm/Group | ARGOS-IO System
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 10/16
Other Adverse Events (participants affected / at risk) | 8/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARGOS-IO System (N=16)
Myocardial infarction (Cardiac disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Increased intraocular pressure (Investigations) | 2 (2)
Increased intraocular pressure -non-study eye- (Investigations) | 1 (1)
Arthralgia -shoulder- (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Plasma cell myeloma in remission (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Loosening of shoulder joint prothesis (Product Issues) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1)
Joint arthroplasty (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARGOS-IO System (N=16)
Visual acuity reduced (Eye disorders) | 3 (3)
Visual acuity reduced -non-study eye- (Eye disorders) | 2 (2)
Reduced general health (General disorders) | 2 (2)
Intraocular pressure increased (Investigations) | 2 (2)
Anterior chamber inflammation (Eye disorders) | 1 (1)
Arthralgia -knee- (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blepharitis (Eye disorders) | 1 (1)
Cardiovascular decompensation (Cardiac disorders) | 1 (1)
Cataract surgery (Surgical and medical procedures) | 1 (1)
Conjunctival irritation b/o allergy to preservatives (Eye disorders) | 1 (1)
Conjunctivitis allergic OU (Eye disorders) | 1 (1)
Conjunctivitis OU (Infections and infestations) | 1 (1)
Contusion -wrist- (Injury, poisoning and procedural complications) | 1 (1)
Corneal dystrophy OU (Eye disorders) | 1 (1)
Corneal endothelial cell loss (Eye disorders) | 1 (1)
Dermatitis allergic -periocular skin- (Skin and subcutaneous tissue disorders) | 1 (1)
Epiretinal membrane (Eye disorders) | 1 (1)
Eye heamatoma (Eye disorders) | 1 (1)
Fatigue (b/o suspected side effects of medications) (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Glaucoma surgery (Surgical and medical procedures) | 1 (1)
Herpes Keratitis OU (Infections and infestations) | 1 (1)
Increased intraocular pressure -non-study eye- (Eye disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Lentodonesis -non-study eye- (Eye disorders) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Oedema peripheral -leg- (General disorders) | 1 (1)
Optic disk haemorrhage (Eye disorders) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1)
Posterior capsule opacification (Eye disorders) | 1 (1)
Posterior capsule opacification -non-study eye- (Eye disorders) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1)
Retinal tear (Eye disorders) | 1 (1)
Skin lesion -wrists and forearms- (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Visual acuity reduced OU (Eye disorders) | 1 (1)
Worsening of allergic reaction to eye drops (Immune system disorders) | 1 (1)
Worsening of glaucoma (Eye disorders) | 1 (1)
Worsening of glaucoma OU (Eye disorders) | 1 (1)
Wound dehiscence -knee- (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT03651336/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT03651336/SAP_001.pdf